CLINICAL TRIAL: NCT04030247
Title: Impact of Plant Sterol Supplement on LDL-C Lowering in Low-to-Moderate Risk South Asian Patients Participating in a Cardiovascular Disease Prevention Program
Brief Title: Impact of Plant Sterol Supplement on LDL-C Lowering in Low-to-Moderate Risk South Asian Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Piper Biosciences, Inc. (Industry)
Responsible Party: Principal Investigator, Rajesh Dash, MD PHD, Director, SSATHI & CardioClick Clinics; Associate Professor of Cardiovascular Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 51046
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Plant Sterol (Experimental): South Asian participants with moderate cardiovascular disease risk will receive standard of care in addition to the plant sterol supplement to take twice daily for 3 months.
  Interventions: Drug: Plant Sterol

INTERVENTIONS:
Drug: Plant Sterol — Patients will receive a plant sterol supplement to take twice daily from their cardiologist/dietician in management of their moderate risk of cardiovascular disease.

SUMMARY:
The purpose of this study is to measure the incremental effectiveness of a twice daily plant sterol supplement in a population of South Asian patients who have low-to-moderate cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
In this study, we aim to measure the LDL-C reducing impact of regular plant sterol supplementation added to a proven CVD reduction program for low-to-moderate risk South Asians who do not meet guideline-based criteria (2018 ACC/AHA Lipid Guidelines) for medical lowering of their LDL-C with an HMG CoA reductase inhibitor (statin) drug, and they are recommended to improve their lipid-risk profile through diet and exercise primarily. In addition, patients who may qualify for statin therapy, but are deemed to be intolerant of statins or who refuse lipid lowering medication may also qualify.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a South Asian male or female, ≥18 years of age
2. Subject has LDL-C ≥120 and <190 mg/dL measured in the past 3 months (or measured at the baseline visit), while not taking cholesterol-lowering medication or cholesterol-lowering supplement for at least 1 month prior, and having a ASCVD Risk score <7.5%.
3. Subjects with LDL-C ≥120 and <190 mg/dL with ASCVD risk scores >7.5% who are known to be intolerant of statin therapy drugs.
4. Subjects with LDL-C > 189 mg/dl or ASCVD > 7.5% who have declined prescription medical therapy.
5. If current smoker, subject does not have any plans to change current smoking status or frequency.
6. Subject is willing to fast (10-14 h, target 12 h, water only) prior to each clinic visit.
7. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.
8. Subject is agreeable to receiving clinical care virtually.

Exclusion Criteria:

1. Subject has taken a prescription cholesterol-lowering medication in the past 1 month.
2. Subject has a known allergy or sensitivity to soy, corn, or other ingredients in the study product.
3. Subject is taking dietary supplements for cholesterol-lowering such as red yeast rice, niacin >100 mg/d or omega-3 fatty acid supplements providing ≥1000 mg/d eicosapentaenoic acid and/or docosahexaenoic acid. (Stable use of viscous fiber laxative ≤2 teaspoons/d is allowed.)
4. Subject is a female, who is pregnant, planning to be pregnant during the study period, or lactating. Subjects should agree to use contraception during study period to avoid pregnancy.
5. Individual has active angina, stable or unstable, requiring urgent cardiovascular functional risk stratification (stress testing or catheterization) or intervention. Or has congestive heart failure that is not compensated or in which the subject is not euvolemic, as determined by the treating MD.
6. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Dash, MD, PhD, Principal Investigator — Stanford University; Gerri O'Riordan, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Plant Sterol: South Asian participants with moderate cardiovascular disease risk receive standard of care in addition to the plant sterol supplement to take twice daily for 3 months.
Period: Overall Study
Arm/Group | Plant Sterol
Started | 50
Completed | 33
Not Completed | 17
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 13

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.33 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 33
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Low Density Lipoprotein-Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 154 (24)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 221 (34)
Calculated LDL-C [Mean (Standard Deviation); unit: mg/dL] | 154 (24)
High Density Lipoprotein-Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 50 (15)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 137 (52)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] — Population: Participants with available data are included in the analysis
  mg/dL
    number analyzed (Participants) | 24
    (all) | 98 (11)
Fasting Insulin [Mean (Standard Deviation); unit: mcU/mL] — Population: Participants with available data are included in the analysis
  mcU/mL
    number analyzed (Participants) | 16
    (all) | 11.3 (7)
Hemoglobin A1C (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin] — Population: Participants with available data are included in the analysis
  Percentage of glycosylated hemoglobin
    number analyzed (Participants) | 22
    (all) | 5.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: LDL-C at Month 3
Time Frame: month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
mg/dL | 145 (20)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.03, t-test, 2 sided

2. Secondary Outcome: Total Cholesterol at Month 3
Time Frame: month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
mg/dL | 216 (29)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.16, t-test, 2 sided

3. Secondary Outcome: Calculated LDL-C at Month 3
Time Frame: month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
mg/dL | 145 (20)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.03, t-test, 2 sided

4. Secondary Outcome: HDL-C at Month 3
Time Frame: month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
mg/dL | 50 (13)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.9, t-test, 2 sided

5. Secondary Outcome: Triglycerides at Month 3
Time Frame: month 3
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 33
mg/dL | 142 (58)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.5, t-test, 2 sided

6. Secondary Outcome: Fasting Glucose at Month 3
Time Frame: month 3
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 24
mg/dL | 96 (8)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.4, t-test, 2 sided

7. Secondary Outcome: Fasting Insulin at Month 3
Time Frame: month 3
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: mcU/mL
Arm/Group | Plant Sterol
Number analyzed (Participants) | 17
mcU/mL | 10.2 (5.9)

8. Secondary Outcome: HbA1c at Month 3
Time Frame: month 3
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | Plant Sterol
Number analyzed (Participants) | 22
Percentage of glycosylated hemoglobin | 5.5 (0.2)
Statistical Analysis 1: Comparison: Plant Sterol; Difference between baseline and month 3; Test type: Other; p = 0.6, t-test, 2 sided

9. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to 3 Months
Description: % change in baseline measurement non-HDL-C to 3 months
Time Frame: Baseline, 3 months
Population: Data were not collected for this outcome measure due to changes in study conduct during the Covid-19 emergency and due to cost of testing that would have been borne by study participants.
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

10. Secondary Outcome: Percent Change in Lp(a) From Baseline to 3 Months
Description: % change in baseline measurement Lp(a) to 3 months
Time Frame: Baseline, 3 months
Population: as for outcome 9
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

11. Secondary Outcome: Percent Change in Apoprotein B-100 From Baseline to 3 Months
Description: % change in baseline measurement Apoprotein B-100 to 3 months
Time Frame: Baseline, 3 months
Population: as for outcome 9
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

12. Secondary Outcome: Percent Change in Apoprotein A1 From Baseline to 3 Months
Description: % change in baseline measurement Apoprotein A1 to 3 months
Time Frame: Baseline, 3 months
Population: as for outcome 9
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

13. Secondary Outcome: Percent Change in Ratio, ApoB-100/Apo A1 From Baseline to 3 Months
Description: % change in baseline measurement ratio, ApoB-100/Apo A1 to 3 months
Time Frame: Baseline, 3 months
Population: as for outcome 9
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

14. Secondary Outcome: Percent Change in C-reactive Protein From Baseline to 3 Months
Description: % change in baseline measurement in C-reactive protein to 3 months
Time Frame: Baseline, 3 months
Population: as for outcome 9
Arm/Group | Plant Sterol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Plant Sterol
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT04030247/Prot_SAP_000.pdf